CLINICAL TRIAL: NCT06038552
Title: Comparison of Clinical Efficacy of Liver Resection, Radiofrequency Ablation, Transarterial Chemoembolization, and Drug Therapy in Patients with Liver Metastasis of Gastrointestinal Stromal Tumors
Brief Title: Comparison of Clinical Efficacy of Liver Resection, RFA, TACE, and Drug Therapy in Patients with GIST LM
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xinhua Zhang, MD, Deputy Director, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: No.[2023]352
Record Dates: First submitted 2023-09-05; First posted 2023-09-15 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: GIST, Malignant; Liver Metastases
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate; Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- IM group: Imatinib(IM)
  Interventions: Drug: imatinib (IM)
- IM combined with HR group: Imatinib(IM) combined with hepatic resection(HR)
  Interventions: Drug: imatinib (IM); Procedure: hepatic resection (HR)
- IM combined with RFA or TACE group: Imatinib(IM) combined with radiofrequency ablation (RFA) or transarterial chemoembolization (TACE)
  Interventions: Drug: imatinib (IM); Procedure: radiofrequency ablation (RFA); Procedure: transarterial chemoembolization (TACE)

INTERVENTIONS:
Drug: imatinib (IM) — Patients with GIST liver metastases were administered an initial IM dose of 400 mg daily, while those with KIT exon 9 mutations received 600-800 mg daily. All patients continued IM indefinitely unless progression or intolerable adverse reactions.
  Other Names: Gleevec
Procedure: hepatic resection (HR) — HR The determination of the surgical modality was established subsequent to comprehensive consultations tailored to each patient within the Department of Liver Surgery. The surgical strategy was established in consideration of factors such as the residual liver volume, tumour positioning, and the surgeon's personal preference. Employing an intraoperative ultrasonographic to enhance the precision of operative assessment.
  Groups: IM combined with HR group
Procedure: radiofrequency ablation (RFA) — RFA RFA was executed utilizing the commercially accessible Cool-tip™ RFA system or the RF 2000 system. The electrode was percutaneously inserted through a guide needle under real-time ultrasound guidance.The primary objective of the RFA procedures encompassed the complete elimination of the tumour entity, with a prescribed ablative margin of 0.5 cm meticulously factored in.
  Groups: IM combined with RFA or TACE group
Procedure: transarterial chemoembolization (TACE) — TACE Under a comprehensive assessment of the hepatic arterial blood supply, a selective catheter was introduced into the segmental or subsegmental arteries that supplied the tumour. The regimen of hepatic arterial infusion chemotherapy included infusion of carboplatin 300 mg, a mixture of 50 mg of epirubicin and 8 mg of mitomycin C, intimately blended with 5 mL of lipiodol. Embolization was finally performed with either absorbable gelatin sponge particles or polyvinyl alcohol particles .
  Groups: IM combined with RFA or TACE group

SUMMARY:
The goal of this observational study is to evaluate the overall survival benefits of local treatment combined with imatinib(IM) and IM alone in patients suffering from GIST liver metastases. The main question it aims to answer is:

• Whether IM combined with hepatic resection (HR) or other local treatments such as radiofrequency ablation (RFA) and transarterial chemoembolization (TACE) has better long-term survival benefits compared to IM monotherapy.

Patients are divided into different treatment groups:

* IM group
* IM combined with HR group
* IM combined with RFA or TACE group

Researchers will compare the IM + HR group and IM + RFA/TACE group with the IM group to see if it has a better Overall survival (OS).

DETAILED DESCRIPTION:
Gastrointestinal stromal tumors (GISTs) represent the most prevalent type of mesenchymal tumor within the gastrointestinal tract, and the liver is the most common site of metastasis from GIST. Imatinib (IM) has significantly enhanced clinical outcomes for patients with advanced disease. Since its approval in February 2002 for treating metastatic or unresectable GISTs, 38% of patients have shown a partial response, while 13.6% have experienced disease progression within 1 to 3 months of IM administration. Over half of the patients with metastases experienced disease progression within two years of IM treatment, attributed to secondary drug resistance. Few studies are comparing the survival benefits of different surgical modalities. The investigators aimed to evaluate IM combined with hepatic resection (HR) or other local treatments such as radiofrequency ablation (RFA) and transarterial chemoembolization (TACE), compared to IM monotherapy in long-term survival benefits in patients suffering from GIST liver metastases.

ELIGIBILITY:
Inclusion Criteria:

* Pathological evidence of GIST of primary tumors
* Liver metastases evidenced by biopsy or radiological findings
* Sufficient liver, hematologic, and renal function, coupled with an Eastern Cooperative Oncology Group performance status score ranging from 0 to 1

Exclusion Criteria:

* IM was not used during treatment
* Liver metastases appeared on second-line or later subsequent lines of TKI
* Combined with other malignant tumors
* Failure to follow up

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2002 to April 2022, 330 consecutive patients were diagnosed with GIST liver metastases. Finally, a total of 238 patients were enrolled in our study. The patients were segregated into different treatment categories: IM therapy (n=126), IM combined with HR (n=81) and IM combined with RFA/TACE (n=31).
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2002-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Overall survival | up to 200 months
  Overall survival (OS) was the span between GIST liver metastases diagnosis and the date of death.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No